CLINICAL TRIAL: NCT01043445
Title: G Protein-coupled Receptor in the Intestine (GPR 119) Stimulated GLP-1 Secretion
Brief Title: -Oleoyl Glycerol is a GPR119 Agonist and Signals GLP-1 Release in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Katrine Bagge Hansen, MD, Ph.d, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GPR119
Record Dates: First submitted 2009-12-02; First posted 2010-01-06 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
Keywords: GPR 119; GLP-1 secretion; 2-oleoyl-glycerol; Dietary supplementation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Oleic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GPR119 agonist, 2-oleoyl glycerol (Experimental): 2-oleoyl glycerol; 2g. and vehicle
  Interventions: Dietary Supplement: GPR 119 agonist, 2-oleyl glycerol; Dietary Supplement: Vehicle
- Oleic acid (Active Comparator): oleic acid; 3.2g and vehicle
  Interventions: Dietary Supplement: Oleic acid; Dietary Supplement: Vehicle
- Vehicle (Placebo Comparator): 5 ml. of glycerol and 5 ml 96% ethanol
  Interventions: Dietary Supplement: Vehicle

INTERVENTIONS:
Dietary Supplement: GPR 119 agonist, 2-oleyl glycerol — Emulgation, 50 ml. containing 2g 2OG
  Arms: GPR119 agonist, 2-oleoyl glycerol
Dietary Supplement: Oleic acid — Emulgation, 50 ml. containing 1.54g of oleic acid
  Arms: Oleic acid
Dietary Supplement: Vehicle — Fifty milliliters of glycerol (Sigma-Aldrich; batch 32296AK, purity 99%) plus 5 ml 96% ethanol

SUMMARY:
The purpose of this study is to evaluate the impact of different ligands of GPR 119 (a G protein-coupled receptor in the intestine) on the secretion of the incretin hormones, GLP-1 and GIP.

DETAILED DESCRIPTION:
We have found a new ligand for the GPR 119 receptor. This study evaluate the impact of this ligand on the incretion hormone responses, beta cell function and gall bladder function in healthy young men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasians v- Normal OGTT (75 g of glucose) according to WHO's criteria
* Normal hemoglobin
* Informed consent

Exclusion Criteria:

* Liver disease (ALAT> 2x normal level)
* Nephropathy (s-creatinin >130 microM or albuminuria)
* Relatives with type 2 diabetes

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The effect of this newly discovered GPR 119 agonist on gut hormone responses, in particular GLP-1 in response of the different meals administered to the subjects | 1 year

SECONDARY OUTCOMES:
Glucose homeostasis, gall bladder contraction in response of the different meals administered to the subjects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Katrine B Hansen, MD, Principal Investigator — Glostrup Hospital, University of Copenhagen; Filip K Knop, MD, Ph.d, Study Director — Gentofte Hospital; Harald S Hansen, professor, Study Director — Farmaceutical Faculty, University of Copenhagen; Jens J Holst, MD;DMSc, Study Director — Biomedical Science, University of Copenhagen
Locations (1):
- Department of Clinical Physiology, Glostrup Hospital, Glostrup Municipality, Denmark